CLINICAL TRIAL: NCT04270201
Title: Determination of ALDH1b1 and ALDH2 Polymorphisms Frequency in the Brazilian Population
Acronym: ALDH2020
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Instituto de Ciências Biomédicas da Universidade de São Paulo (Unknown)
Responsible Party: Sponsor
Other Study IDs: NP1553/19
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Oral Squamous Cell Carcinoma (OSCC)
Keywords: Oral squamous cell carcinoma; ALDH1b1; ALDH2; polymorphism
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: OSCC patients (n = 60)
  Interventions: Other: Saliva collection
- Control group: Healthy volunteers (n = 240)
  Interventions: Other: Saliva collection

INTERVENTIONS:
Other: Saliva collection — Saliva collection

SUMMARY:
A case-control study with oral squamous cell carcinoma (OSCC) patients from Instituto do Câncer do Estado de São Paulo (ICESP) and healthy volunteers. In this study, it will be collected saliva samples from both groups that will be submitted to sequencing analysis to evaluate the frequency of ALDH1b1 and ALDH2 polymorphisms in the Brazilian population. Also, correlate OSCC risk to alcohol consumption or smoke, by applied questionnaires.

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), in 2016 there were 3 million deaths worldwide from alcohol abuse. ALDH1b1 and ALDH2 proteins are involved in the alcohol metabolism promoting the conversion of acetaldehyde to acetate. The genes that encode these proteins have genetic variants, also called polymorphisms, that can promote changes in their functions such as the accumulation of acetaldehyde in the body, resulting in facial flushing, tachycardia and headache. Studies reported the correlation between alcohol consumption and/or smoking and these polymorphisms to a higher risk for head and neck cancer, including oral squamous cell carcinoma (OSCC). The aim of this study is to determine the frequency of the ALDH1b1 and ALDH2 polymorphisms in the Brazilian population, in addition to estimating the risk for OSCC among those with polymorphisms. For this, unstimulated saliva samples will be collected from OSCC patients and healthy volunteers. All study participants must complete two questionnaires on alcohol consumption, smoking and disease history. Saliva samples will be collected using the DNA/RNA Shield Saliva Collection Kit and stored at -20ºC. The DNA will be extracted, quantified by the Nanodrop equipment and amplified by the polymerase chain reaction (PCR), using specific primers for each of the genetic variants. The PCR product will be sent to the Sequencing Service of the Centro de Pesquisas sobre o Genoma Humano e Células-Tronco/IBUSP, where the Sanger sequencing technique will be performed and the results will be analyzed in the ICB-USP laboratory. For the group of patients, medical records will be monitored to correlate clinical data and genetic variants with overall survival. These data will allow the characterization of the genetic variants of ALDH1b1 and ALDH2 in the Brazilian population and support the development of future public policies to reduce the main risk factors for OSCC, especially among those with these genetic variants.

ELIGIBILITY:
Inclusion Criteria:

* OSCC diagnostic for case group
* Able to read and sign the consent form.
* Able for saliva collection.
* Able to understand the applied questionnaires.

Exclusion Criteria:

* Unable to read and sign the consent form.
* Unable for saliva collection.
* Unable to understand the applied questionnaires.
* OSCC patient's companions for healthy volunteers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OSCC patients (n = 60) and healthy volunteers (n = 240) matched by age and sex.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-02 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of ALDH1b1 and ALDH2 polymorphisms | 1 year
  Determine the frequency of ALDH1b1 and ALDH2 polymorphisms in OSCC patients and healthy volunteers.

SECONDARY OUTCOMES:
Survival | 5 years
  Overall survival (case group)

CONTACTS AND LOCATIONS:
Overall Officials: Gilberto de Castro Junior, MD, PhD, Principal Investigator — Instituto do Câncer do Estado de São Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil